CLINICAL TRIAL: NCT06376435
Title: A Multicentre Real-world Study of Heptapopal Ethanolamine Tablets in Concurrent/Sequential Radioimmunoinduced Thrombocytopenia
Status: Not yet recruiting | Type: Observational
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Principal Investigator, Jun wang, study principal investigator, Hebei Medical University Fourth Hospital
Other Study IDs: HBHQ-CTIT-RWS
Record Dates: First submitted 2024-04-11; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Cancer, Therapy-Related
MeSH Terms: conditions — Neoplasms, Second Primary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Single drug group
  Interventions: Drug: Herombopag Olamine Tablets
- combined rhTPO group
  Interventions: Drug: Herombopag Olamine Tablets
- combined IL-11 group
  Interventions: Drug: Herombopag Olamine Tablets

INTERVENTIONS:
Drug: Herombopag Olamine Tablets — Herombopag Olamine；combined rhTPO;combined IL-11

SUMMARY:
The objective of this study was to observe and evaluate the efficacy and safety of hexapopal ethanolamine tablets in the treatment of synchronous/sequential radioimmunoinduced thrombocytopenia in the real world.

The subjects of this study were patients with solid malignant tumors who had received radioimmunoinduced thrombocytopenia.

This study will retrospectively and prospectively collect real-world data related to investigational drugs, and will observe 500 patients to observe the diagnosis and treatment pattern of radiochemo-induced thrombocytopenia. The study included a screening period (no more than one week) and a treatment period (at least two cycles).Participants meeting protocol inclusion criteria were defined as having platelet values < 100×109/L during radioimmunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Understand the research procedure and voluntarily sign the informed consent to participate in the study
* Subjects ≥18 years of age receiving synchronous/sequential chemotherapeutic therapy
* Patients with platelet count ≤100×109/L or platelet count decrease ≥ 50×109/L or platelet count > 100×109/L but need to be prophylaxis with hexapopethanolamine tablets
* Researchers believe that subjects need to be treated with hexapopal.

Exclusion Criteria:

* The subjects are conducting clinical intervention studies
* Patients with known or expected allergy or intolerance to the active ingredient or excipient of hexapopar
* Pregnant or lactating women
* Other conditions deemed unsuitable for inclusion in the study by the researcher.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with solid malignancies undergoing radiotherapy/chemotherapy/immunosuppressant induced thrombocytopenia
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-04-20 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients recovered to 100×109/L | 14 days after starting treatment with the study drug
  The proportion of patients who recovered to 100×109/L within 14 days after starting treatment with the drug was studied

SECONDARY OUTCOMES:
The proportion of patients recovered to 75×109/L | up to 2 months
  The proportion of patients who recovered to 75×109/L after starting treatment with the drug was studied
Time for platelet recovery to 100×109/L | up to 2 months
  Study the time for platelet recovery to 100×109/L after drug initiation
Proportion of patients with treatment delay or dose reduction | up to 2 months
  Proportion of patients with delayed or reduced dose of radiotherapy, chemotherapy, immunosuppressants, etc
TRAE | up to 2 months
  Study drug-related adverse reactions